CLINICAL TRIAL: NCT03868722
Title: Short-term Combined Acalabrutinib and Venetoclax Treatment of Newly Diagnosed Patients With CLL at High Risk of Infection and/or Early Treatment, Who do Not Fulfil IWCLL Treatment Criteria.
Brief Title: Acalabrutinib and Venetoclax Treatment of Newly Diagnosed Patients With CLL at High Risk of Infection or Early Treatment
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Carsten Utoft Niemann, MD, PhD, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PreVent-ACaLL
Record Dates: First submitted 2019-02-26; First posted 2019-03-11 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: CLL
MeSH Terms: interventions — acalabrutinib; venetoclax

STUDY DESIGN:
Intervention Model Description: Randomization has to occur within 42 days after the first tests for screening were performed. Patients will be randomly assigned to treatment vs observation through 1:1 randomization process with stratification according to country, TP53 aberration status and IGHV mutational status. Treatment or observation period has to be initiated within 14 days after randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Experimental): Treatment with Acalabrutinib and Venetoclax is initiated within 14 days after randomization.
  Interventions: Drug: Acalabrutinib; Drug: Venetoclax
- Observation arm (No Intervention): Observation period is initiated within 14 days after randomization.

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib 100 mg BID from cycle 1 day 1 for 3 cycles of 28 days.
  Other Names: Calquence
  Arms: Treatment arm
Drug: Venetoclax — Venetoclax, ramp up during the first five weeks starting cycle 1 day 1, 7 days treatment on each dose level (20-50-100-200-400 mg), thereafter 400 mg once daily for a total of 3 cycles of 28 days.
  Other Names: Venclexta; Venclyxto
  Arms: Treatment arm

SUMMARY:
Many patients with CLL have a weakened immune system due to their disease. It increases their risk of developing serious, treatment-requiring infections such as blood poisoning or pneumonia, which in the worst case may end with fatal outcomes.

Serious infections due to CLL are responsible for one third of all deaths among CLL patients. PreVent-ACaLL study will investigate whether a combination of two known types of cancer drugs can reduce the risk of infection and thus mortality when given preventively to newly diagnosed CLL patients.

A newly developed register-based computer model can predict which patients are at high risk in order to develop infections as a result of their CLL. A preventive treatment might be initiated before patients need chemotherapy. In this way, the cancer disease might be "reset" so that the immune system, which is inhibited by CLL, is restored and the risk of fatal infections is minimized.

DETAILED DESCRIPTION:
OBJECTIVE AND HYPOTHESIS Phase 2, randomized study of short-term, combined venetoclax and acalabrutinib treatment of newly diagnosed patients with CLL. For patients identified by CLL-TIM (the Machine Learning predictive algorithm, Treatment Infection Model) at high risk of infection and/or early CLL treatment, it is tested whether grade 3-Infection-free, treatment-free survival can be improved by three months of venetoclax+acalabrutinib treatment. Changes in immune dysfunction are measured by an extensive translational program for correlation with changes in infection.

BACKGROUND Infection and immune dysfunction in patients diagnosed with CLL leads to significant morbidity and mortality, as exemplified by the constant rate of infectious deaths in CLL over the last three decades, despite significant improvement in all other causes of death. This also affects patients who do not need treatment according to IWCLL criteria, thus infections are the leading cause of death among patients with CLL. Based on a novel machine learning algorithm, CLL-TIM, patients at high risk (>65% 2-years risk) of severe infection and/or CLL treatment can be identified at diagnosis. By a short period of preemptive treatment for these patients, the aim is to change the natural history of CLL and immune dysfunction.

METHODS The study is an intergroup study between the HOVON (Belgium, the Netherlands) and the Nordic (Denmark, Norway, Sweden, Finland) CLL study groups. For the phase 2 study, 4-8 sites with the capacity of the extensive translational immune phenotyping and/or timely shipment of samples will be selected. Patients are randomized between venetoclax+acalabrutinib treatment for three months or observation. For each treatment arm, 25 patients are needed (50 in total). Thorough assessment of immune function before, during and after treatment as well as detailed reporting on infectious complications, the proof of concept of the PreVent-ACaLL study's capacity to change the natural history of immune dysfunction in CLL by short-term venetoclax-acalabrutinib treatment will be made.

PERSPECTIVES By addressing the unmet need of improving immune function for newly diagnosed CLL patients with high risk of infections and/or early CLL treatment, the aim is to change the paradigm for CLL treatment and the natural history of the disease.

If the phase 2 trial demonstrates a clear signal for safety with indication of benefit for patients in the treatment arm, an extension phase 3 study is planned with the potential to change the future management of CLL.

ELIGIBILITY:
Inclusion Criteria:

1. CLL diagnosed according to IWCLL criteria within one year prior to randomization
2. High risk of infection and/or progressive treatment within 2 years according to CLL-TIM
3. IWCLL treatment indication not fulfilled
4. Life expectancy > 2 years
5. Age at least 18 years
6. Ability and willingness to provide written informed consent and adhere to study procedures and treatment
7. Adequate bone marrow function as indicated by platelets above 100 x 10E9, hemoglobin above 10 g/dL and neutrophils above 1 x 10E9
8. Creatinine clearance above 30 mL/min directly measured with 24hr urine collection or calculated according to the modified formula of Cockcroft and Gault
9. Adequate liver function as indicated by a total bilirubin≤ 2 x, AST/ALT ≤ 2.5 x the institutional ULN value, unless directly attributable to the patient's CLL or to Gilbert's Syndrome.
10. Negative serological testing for hepatitis B (HBsAg negative and anti-HBc negative; patients positive for anti-HBc may be included if PCR for HBV DNA is negative and HBV-DNA PCR is performed every month until 12 months after last treatment cycle), negative testing for hepatitis C RNA within 6 weeks prior to registration.
11. Eastern Cooperative Oncology Group Performance Status (ECOG) performance status 0-2.
12. Woman of childbearing potential (WOCBP) who are sexually active must use highly effective methods of contraception during treatment and for 2 days after the last dose of investigational drugs.
13. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty.
14. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information

Exclusion Criteria:

1. Prior CLL treatment (including monoclonal antibodies, chemotherapy, small molecules)
2. Transformation of CLL (Richter's transformation)
3. Previous autoimmune disease as AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura) treated with immune suppression or uncontrolled AIHA or ITP
4. History of PML
5. Uncontrolled or active infection
6. Malignancies other than CLL requiring systemic therapies (except anti-hormonal therapies) or considered to impact survival
7. Requirement of therapy with strong CYP3A4 and CYP3A5 inhibitors/inducers or anticoagulant therapy with vitamin K antagonists
8. History of bleeding disorders or current platelet inhibitors or anticoagulant therapy
9. History of clinically significant cardiovascular disease such as arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or corrected QT interval (QTc) > 480 msec at screening.
10. History of stroke or intracranial hemorrhage within 6 months prior to registration.
11. Use of investigational agents which might interfere with the study drug within 28 days prior to registration.
12. Vaccination with live vaccines 28 days prior to registration.
13. Major surgery less than 30 days before start of treatment.
14. Known hypersensitivity to any active substance or to any of the excipients of one of the drugs used in the trial.
15. Pregnant women and nursing mothers (a negative pregnancy test is required for all women of childbearing potential within 7 days before start of treatment; further pregnancy testing will be performed regularly).
16. Fertile men or women of childbearing potential unless: surgically sterile or ≥ 2 years after the onset of menopause or willing to use two methods of reliable contraception including one highly effective contraceptive method (Pearl Index <1) and one additional effective (barrier) method during study treatment and for 18 months after the end of study treatment.
17. Legal incapacity.
18. Persons who are in dependence to the sponsor or an investigator
19. Persons not considered fit for the trial by the investigator
20. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
21. Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening.
22. Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer.
23. Prothrombin time/INR or aPTT (in the absence of Lupus anticoagulant) > 2x ULN.
24. Requires treatment with proton pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
25. Major surgical procedure within 7 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
26. Breastfeeding or pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2019-10-11 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Grade 3-Infection-free survival | 12 weeks after finishing treatment
  Grade 3-Infection-free survival in the treatment arm compared to the observation arm
Event-free survival | 2 years after enrollment
  Event-free survival, event being either grade ≥3 infection or CLL treatment

SECONDARY OUTCOMES:
Event-free survival | 12 weeks after treatment initiation,1 year and 2 years after enrollment
  Event-free survival, event being either grade ≥3 infection or CLL treatment
Overall survival | Assessed at 12 weeks, 1 year and 2 years from treatment/observation initiation
  Overall survival
Treatment free survival | Assessed at 12 weeks, 1 year and 2 years from treatment/observation initiation
  Treatment free survival
Rate of infections | assessed at 12 weeks, 1 year and 2 years from treatment/observation initiation
  Rate of infections
Rate of infections grade ≥3 | assessed at 12 weeks, 1 year and 2 years from treatment/observation initiation
  Rate of infections

CONTACTS AND LOCATIONS:
Overall Officials: Carsten U Niemann, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (7):
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - Herlev og Gentofte Hospital, Herlev
  - Sjællands Universitetshospital Roskilde, Roskilde
- Netherlands (2):
  - Albert Schweitzer Hospital, Dordrecht
  - Ikazia Hospital (Ikazia Ziekenhuis), Rotterdam
- Sweden (2):
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No
Restricted access based on individual agreements based on Danish and EU legislation

REFERENCES:
- [Background] Barf T, Covey T, Izumi R, van de Kar B, Gulrajani M, van Lith B, van Hoek M, de Zwart E, Mittag D, Demont D, Verkaik S, Krantz F, Pearson PG, Ulrich R, Kaptein A. Acalabrutinib (ACP-196): A Covalent Bruton Tyrosine Kinase Inhibitor with a Differentiated Selectivity and In Vivo Potency Profile. J Pharmacol Exp Ther. 2017 Nov;363(2):240-252. doi: 10.1124/jpet.117.242909. Epub 2017 Sep 7. PMID 28882879
- [Background] Bradshaw JM. The Src, Syk, and Tec family kinases: distinct types of molecular switches. Cell Signal. 2010 Aug;22(8):1175-84. doi: 10.1016/j.cellsig.2010.03.001. Epub 2010 Mar 4. PMID 20206686
- [Background] de Rooij MF, Kuil A, Geest CR, Eldering E, Chang BY, Buggy JJ, Pals ST, Spaargaren M. The clinically active BTK inhibitor PCI-32765 targets B-cell receptor- and chemokine-controlled adhesion and migration in chronic lymphocytic leukemia. Blood. 2012 Mar 15;119(11):2590-4. doi: 10.1182/blood-2011-11-390989. Epub 2012 Jan 25. PMID 22279054
- [Background] Khan WN. Regulation of B lymphocyte development and activation by Bruton's tyrosine kinase. Immunol Res. 2001;23(2-3):147-56. doi: 10.1385/IR:23:2-3:147. PMID 11444380
- [Background] Mohamed AJ, Yu L, Backesjo CM, Vargas L, Faryal R, Aints A, Christensson B, Berglof A, Vihinen M, Nore BF, Smith CI. Bruton's tyrosine kinase (Btk): function, regulation, and transformation with special emphasis on the PH domain. Immunol Rev. 2009 Mar;228(1):58-73. doi: 10.1111/j.1600-065X.2008.00741.x. PMID 19290921
- [Background] Ponader S, Chen SS, Buggy JJ, Balakrishnan K, Gandhi V, Wierda WG, Keating MJ, O'Brien S, Chiorazzi N, Burger JA. The Bruton tyrosine kinase inhibitor PCI-32765 thwarts chronic lymphocytic leukemia cell survival and tissue homing in vitro and in vivo. Blood. 2012 Feb 2;119(5):1182-9. doi: 10.1182/blood-2011-10-386417. Epub 2011 Dec 16. PMID 22180443
- [Background] Smith TJ, Khatcheressian J, Lyman GH, Ozer H, Armitage JO, Balducci L, Bennett CL, Cantor SB, Crawford J, Cross SJ, Demetri G, Desch CE, Pizzo PA, Schiffer CA, Schwartzberg L, Somerfield MR, Somlo G, Wade JC, Wade JL, Winn RJ, Wozniak AJ, Wolff AC. 2006 update of recommendations for the use of white blood cell growth factors: an evidence-based clinical practice guideline. J Clin Oncol. 2006 Jul 1;24(19):3187-205. doi: 10.1200/JCO.2006.06.4451. Epub 2006 May 8. PMID 16682719
- [Background] Soucek L, Buggy JJ, Kortlever R, Adimoolam S, Monclus HA, Allende MT, Swigart LB, Evan GI. Modeling pharmacological inhibition of mast cell degranulation as a therapy for insulinoma. Neoplasia. 2011 Nov;13(11):1093-100. doi: 10.1593/neo.11980. PMID 22131884
- [Derived] Svanberg Teglgaard R, Marquart HV, Hartling HJ, Bay JT, da Cunha-Bang C, Brieghel C, Faitova T, Enggaard L, Kater AP, Levin MD, Kersting S, Ostrowski SR, Niemann CU. Improved Innate Immune Function in Patients with Chronic Lymphocytic Leukemia Treated with Targeted Therapy in Clinical Trials. Clin Cancer Res. 2024 May 1;30(9):1959-1971. doi: 10.1158/1078-0432.CCR-23-2522. PMID 38393694
- [Derived] Gargiulo E, Teglgaard RS, Faitova T, Niemann CU. Immune Dysfunction and Infection - Interaction between CLL and Treatment: A Reflection on Current Treatment Paradigms and Unmet Needs. Acta Haematol. 2024;147(1):84-98. doi: 10.1159/000533234. Epub 2023 Jul 27. PMID 37497921